CLINICAL TRIAL: NCT01054014
Title: A Double-Blind, Placebo-Controlled, Randomized, Single and Multiple Ascending Dose Study to Investigate the Safety, Tolerability, Food Effect, and Pharmacokinetics of JNJ-40346527 in Healthy Subjects
Brief Title: A Single and Multiple Dose Study to Explore the Safety Of JNJ-40346527 In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR016795
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Health
Keywords: CR016795
MeSH Terms: interventions — JNJ-40346527

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 001 (Experimental): JNJ-40346527/Placebo Single oral dose of JNJ-40346527 (either 10 50 150 300 600 or 1000mg) or Placebo
  Interventions: Drug: JNJ-40346527/Placebo
- 002 (Experimental): JNJ-40346527/Placebo JNJ-40346527 once daily oral dose for 14 days (either 50 150 300 500 or 750mg) or Placebo
  Interventions: Drug: JNJ-40346527/Placebo
- 003 (Experimental): JNJ-40346527 JNJ-40346527 150mg one dose either fasting (or with food) then after 7 days off treatment JNJ-40346527 150mg either with food (or fasting)
  Interventions: Drug: JNJ-40346527

INTERVENTIONS:
Drug: JNJ-40346527/Placebo — Single oral dose of JNJ-40346527 (either 10, 50, 150, 300, 600, or 1000mg) or Placebo
  Arms: 001
Drug: JNJ-40346527/Placebo — JNJ-40346527 once daily oral dose for 14 days (either 50, 150, 300, 500 or 750mg) or Placebo
  Arms: 002
Drug: JNJ-40346527 — JNJ-40346527 150mg one dose, either fasting (or with food), then after 7 days off treatment, JNJ-40346527 150mg either with food (or fasting)
  Arms: 003

SUMMARY:
The purpose of this study is to investigate the safety, tolerability and pharmacokinetics (how the drug is absorbed in the body, how it is distributed within the body and it is removed from the body over time) of single and multiple doses of JNJ-40346527 in healthy volunteers. This study will also investigate the pharmacokinetics of JNJ-40346527 with and without food.

DETAILED DESCRIPTION:
JNJ-40346527 is an experimental drug that is being tested to see if it may be useful in treating of rheumatoid arthritis and other inflammatory diseases. This study will compare the effects (both good and bad) of JNJ-40346527 to those of placebo (which looks like the drug being studied but has no active ingredients) in healthy volunteers. This study will be the first study in which JNJ-40346527 is given to humans. This study is being conducted in three parts. Parts 1 and 2 are randomized (study drug will be assigned by chance), double-blind (neither the physician nor volunteer knows the identity of the assigned drug) studies comparing the safety and tolerability of JNJ-40346527 to placebo in 96 healthy volunteers. Part 3 is an open-label (all people involved know the identity of the assigned drug), 2-period crossover (meaning that volunteers will receive both treatments at different times) study of the effects of food on JNJ-40346527 in 8 healthy male volunteers. For Part 1, the participation period is a maximum of 64 days, including a screening visit, a 5-day in-clinic period and three follow-up visits. For Part 2, the participation period is a maximum of 83 days, including a screening visit, an 18-day in-clinic period and two follow-up visits. For Part 3, the participation period is a maximum of 59 days, including a screening visit, two 4-day in-clinic periods separated by a 7 day break, and a follow-up visit. For all three parts of the study, safety evaluations, which will include ECG (a cardiac function test), vital signs and monitoring of side-effects will be performed. Additionally, blood and urine samples will be collected for evaluation. Volunteers will participate in 1 of 3 parts; Part 1: volunteers will receive a single oral (by mouth) dose of JNJ-40346527 (10, 50, 150, 300, 600, or 1000mg) or placebo; Part 2: volunteers will receive oral doses of JNJ-40346527 (50, 150, 300, 500 or 750mg) or placebo once a day for 14 days; Part 3: volunteers will receive two oral doses of 150mg of JNJ-40346527 with and without food, with a 7-day break between doses.

ELIGIBILITY:
Inclusion Criteria:

* Must be generally in good health
* Have negative result for HIV,hepatitis B, and hepatitis C
* Non-smoker for at least 6 months
* Females must be of non childbearing potential,i.e., either: surgically sterile (bilateral tubal ligation or removal of ovaries and/or uterus or partial hysterectomy at least 6 months prior to dosing), or naturally postmenopausal for at least 2 years, with negative blood and urine pregnancy tests prior to dosing
* must consent to use a medically acceptable method of contraception throughout the entire study period and for 90 days after the study is completed

Exclusion Criteria:

* History of alcohol or drug abuse
* Average consumption of more than 5 cups of caffeinated beverages (tea/coffee/cocoa/cola) per day
* History of any type of significant allergies (eg, anaphylaxis, prominent respiratory and skin symptoms)
* Use of St.John's Wort (hypericin) for 30 days before first dosing
* Use of any type of hormone replacement therapy for 30 days before the first dose
* history of receiving a live virus vaccination within the past month or plans to receive vaccination with a live virus vaccine within 2 weeks following the last dose of medication
* receipt of an experimental drug or medical device within the last month

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2010-01; Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To assess the safety, tolerability and pharmacokinetics (PK) of JNJ-40346427 after administration of single and multiple oral ascending doses of JNJ-40346427 in healthy volunteers and the PK of JNJ-4034627 with and without food. | from time of dosing to follow-up (28-35 days)

SECONDARY OUTCOMES:
To assess the pharmacodynamics (explores what the drug does to the body) of JNJ-40346527. | Part 1: Days 1 & 2; Part 2: Days 1, 7, 14, and 15

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Antwerp, Belgium